CLINICAL TRIAL: NCT00725036
Title: A 24-month Multicentre, Open-label, Randomised, Parallel Group, Long Term Safety Trial Comparing Intensive Treatment of Pulmonary Inhaled Human Insulin With Insulin Aspart Administered s.c., Both in Combination With NPH, in Subjects With Type 1 Diabetes
Brief Title: Long Term Safety Trial to Compare Insulin Treatment With Preprandial Inhaled Human Insulin to s.c. Insulin Aspart Both Combined With NPH in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1998-1496
Record Dates: First submitted 2008-07-29; First posted 2008-07-30 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: inhaled human insulin
Drug: insulin aspart
Drug: insulin NPH

SUMMARY:
This trial is conducted in Oceania.

The aim of this trial is to compare the safety of using pulmonary inhaled human insulin to s.c. insulin aspart both combined with NPH insulin in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Current treatment with any insulin in any regimen
* Body mass index (BMI) below 38.0 kg/m2
* HbA1c below or equal to 13.0%

Exclusion Criteria:

* Total daily insulin dosage more than 100 IU/day
* Current acute or chronic pulmonary disease (excluding asthma)
* Recurrent major hypoglycaemia
* Proliferative retinopathy or maculopathy requiring acute treatment
* Smoker
* Chest X-ray with clinically significant abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2002-09-02 (Actual); Primary Completion 2004-12-14 (Actual); Study Completion 2004-12-14 (Actual)

PRIMARY OUTCOMES:
Long term pulmonary safety profiles | during treatment

SECONDARY OUTCOMES:
Glycaemic control as measured by HbA1c
Incidence of hypoglycaemic episodes
Long-term safety profiles (laboratory, ECG, insulin antibodies)
Physical examination and body weight and vital signs
Adverse events
Treatment satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (18):
- Australia (18):
  - Novo Nordisk Investigational Site, Broadmeadow, New South Wales
  - Novo Nordisk Investigational Site, Camperdown, New South Wales
  - Novo Nordisk Investigational Site, St Leonards, New South Wales
  - Novo Nordisk Investigational Site, Wollongong, New South Wales
  - Novo Nordisk Investigational Site, Woolloongabba, Queensland
  - Novo Nordisk Investigational Site, Keswick, South Australia
  - Novo Nordisk Investigational Site, Fremantle, Western Australia
  - Novo Nordisk Investigational Site, Ashford
  - Novo Nordisk Investigational Site, Auckland
  - Novo Nordisk Investigational Site, Box Hill
  - Novo Nordisk Investigational Site, Christchurch
  - Novo Nordisk Investigational Site, Clayton
  - Novo Nordisk Investigational Site, Garran
  - Novo Nordisk Investigational Site, Heidelberg
  - Novo Nordisk Investigational Site, Parkville
  - Novo Nordisk Investigational Site, Perth
  - Novo Nordisk Investigational Site, Randwick
  - Novo Nordisk Investigational Site, Stones Corner

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com